CLINICAL TRIAL: NCT01021891
Title: A Phase 1b, Single-Dose, Open-Label, Parallel, Controlled Pharmacology Trial of Inhaled Technosphere®/Insulin in Non-Diabetic Subjects With COPD Versus Matched Non-Diabetic Subjects Without COPD.
Brief Title: A Study to Evaluate Insulin in the Blood After Inhalation of a Dry Powder Insulin Formulation (Called Technosphere®/Insulin) in Non-diabetic Patients With & Without Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mannkind Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MKC-TI-015; EudraCT Number: 2007-002818-19
Record Dates: First submitted 2009-11-25; First posted 2009-11-30 (Estimated); Last update posted 2013-12-17 (Estimated); Status verified 2013-12

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: Technosphere® Insulin Inhalation Powder
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Non-Diabetic Subj. w/o COPD (Experimental): Single dose, 30 units
  Interventions: Drug: Technosphere®/Insulin
- Non-Diabetic Subj. with COPD (Experimental): Single dose, 30 units
  Interventions: Drug: Technosphere®/Insulin

INTERVENTIONS:
Drug: Technosphere®/Insulin

SUMMARY:
Trial will include 40 subjects and consists of 3 visits: Screening, Treatment and Follow up. A euglycemic clamp procedure and Technosphere®/Insulin (T/I) administration will occur at Visit 2 for both COPD and non COPD subjects.

DETAILED DESCRIPTION:
Trial objectives are to evaluate the impact of a defined lung disease (COPD) on pharmacokinetic parameters of insulin and fumaryl diketopiperazine (FDKP) after inhalation of Technosphere®/Insulin (T/I), the investigational medicinal product. 40 non diabetic subjects, 20 COPD and 20 age/gender/BMI-matched non COPD subjects will participate in 3 visits: Visit 1 (screening), Visit 2 (subjects will undergo a euglycemic clamp procedure and be dosed with T/I) and Visit 3 (follow up visit).

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects minimum 18 and maximum 70 years of age
* Body Mass Index (BMI) = 36 kg/m2
* Subjects with COPD: Diagnosis of COPD (emphysema and/or chronic bronchitis),
* smoking history =10 years, chronic cough present intermittently or daily with or without sputum and/or dyspnea upon exertion.
* Subjects with COPD: Pulmonary Function Tests - FEV1 =50% (NHANES) III
* Predicted; FEV1/FVC < 70 % (NHANES) III; TLC =80% of Predicted (ITS) and DLco(unc) =50% of Predicted (Miller)
* Subjects without COPD: PFTs: FEV1 = 70% NHANES III Predicted; TLC =80% of
* Predicted (ITS) and DLco(unc) =80% of Predicted (Miller)

Exclusion Criteria:

* History of pre-diabetes or diabetes
* Previous or current treatment with any anti-diabetic drugs
* Serum creatinine > 2.0 mg/dL in males and > 1.8 mg/dL in females
* Active smokers defined as having smoked their last cigarette, pipe, and/or cigar without the previous 6 months
* Previous exposure to any inhaled insulin product or investigational medicines/devices within the previous 30 days prior to entry or participation
* Clinically significant major organ disease
* Female subjects of childbearing potential not practicing adequate birth control
* Subjects with COPD: Significant improvement in pre-to post-bronchodilator spirometry (defined as an increase of 12% AND 200 mL in either FVC or FEV1);
* Any clinically important pulmonary disease except mild or moderate COPD
* Subjects without COPD: Any important pulmonary disease confirmed by pulmonary function testing and/or radiologic findings

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2006-07; Primary Completion 2008-08 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
To evaluate the pharmacokinetic disposition of serum insulin and serum fumaryl diketopiperazine following dosing with 30 U T/I, as measured via Area Under the Curve serum insulin and AUC 0-480 min serum FDKP | 30 days

SECONDARY OUTCOMES:
Efficacy endpoints include: additional PK parameters of serum insulin and serum FDKP, Pharmacodynamic parameters of sersum insulin, safety of T/I | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Anders Boss, MD, Study Chair — MannKind Corp
Locations (5):
- Diabetes & Glandular Disease Research Assoc PA, San Antonio, Texas, United States
- Medical University Graz, Graz, Graz, Austria
- University Medical Centre Groningen, Zuidlaren, Netherlands
- United Kingdom (2):
  - Medicines Evaluation Unit (MEU), Manchester, England
  - ICON Development Solutions, Manchester